CLINICAL TRIAL: NCT07332819
Title: Efficacy and Safety of Resveratol I Pediatric and Adolescence With Type 1 Diabetic Nephropathy: A Six Months Preliminary Exploratory Trial
Brief Title: Resveratol in Diabetic Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran yousef, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS 385/2021
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetic Nephropathy
Keywords: Resveratol; Type 1 diabetes; Nephropathy; Children and adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratol (Experimental)
  Interventions: Dietary Supplement: Resveratol
- Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratol — Resveratol oral supplementation
  Arms: Resveratol
Other: Placebo — Oral placebo
  Arms: Control

SUMMARY:
Background: Food-derived compounds have been shown to have beneficial effects in type 1 diabetes mellitus (T1DM). Among these compounds, resveratrol (3,5,4'-trihydroxystilbene) which is found in grapes, peanuts, cranberries. Resveratrol has a wide range of effects including antimicrobial, anti-inflammatory, anti-apoptotic, anticancer, anti-oxidative and cardio- protective effects. Resveratrol is capable of inducing beneficial effects in diabetic animals and thereby, ameliorates diabetes. Recently, resveratrol showed beneficial effects in adults with T1DM. Objectives: Therefore, we performed a randomized-controlled trial to assess the effect of oral resveratrol supplementation on glycemic control, lipid profile and kidney injury molecule-1 (KIM-1) levels in pediatric patients with T1DM and diabetic nephropathy. Methods: This study included 60 children and adolescents with T1DM. Enrolled patients aged 12-18 years with disease duration > 5 years and have diabetic nephropathy. Patients were randomly assigned into two groups; intervention group (group A) who received oral resveratrol tablets 250 mg twice daily. The other group (group B) did not receive any supplementation and served as a control group. Both groups were followed-up for 6 months with assessment of fasting blood glucose (FBG), HbA1c, urinary albumin creatinine ratio (UACR) and KIM-1 levels. Insulin sensitivity score and estimated glucose disposal rate (eGDR) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients with T1DM. 2- Patients aged 12-18 years with at least 5 years disease duration. 3- Active diabetic nephropathy in the form of microalbuminuria (urinary albumin excretion [UAE] 30-299 mg/g creatinine). The presence of persistent microalbuminuria was confirmed by finding two or all of three samples abnormal over a 3- to 6-months period prior to study despite angiotensin converting enzyme inhibitors (ACE-Is) (Tabaei et al., 2001; Molitch et al., 2004; Donaghueet al., 2018). 4- Hemoglobin A1c (HbA1c) ≤9.0%. 5- Patients on regular visit to clinic. 6- Patients on regular insulin therapy.

Exclusion Criteria:

* Patients with history of liver disease or any disorder likely to impair liver functions or elevated liver enzymes (aminotransferases levels higher than twice the upper normal limit). 2. Patients with renal impairment due to cause other than diabetes. 3. Patients with hypertension. 4. Hyper- or hypo-thyroidism. 5. Hepatitis virus infection (B or C) or any evidence of infection. 6. Hypoglycaemic unawareness or recurrent severe hypoglycaemic episode in 6 months prior to recruitment. 7. Recurrent diabetic ketoacidosis (more than 2 episodes in the previous 12 months). 8. Serious co-morbidities. 9. Patients were already on anti-hypertensive drugs or any antioxidant therapy such as vitamin supplements. 10. Taking any vitamins or food supplements one month before study. 11. Patients who have an allergy to grapes, berries, and peanuts. 12. Participation in a previous investigational drug study within 3 months preceding screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-21 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Improvement in time in range at the study endpoint. | 6 months.

SECONDARY OUTCOMES:
Change in serum KIM-1 measured by Elisa at the study endpoint. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No